CLINICAL TRIAL: NCT06663904
Title: Multicenter Validation of Different Abbreviated MRI Protocols for Early-Stage Hepatocellular Carcinoma Diagnosis Using Main and Ancillary Features of LI-RADS
Brief Title: Different Abbreviated MRI for Hepatocellular Carcinoma Diagnosis
Acronym: AMRI; LIRADS
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yanjin Qin, clinical doctor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: SYSUFAH2021124; 82271958 (Other Grant/Funding Number: National Natural Science Foundation of China); 2024A1515012149, 2023A15150110 (Other Grant/Funding Number: Natural Science Foundation of Guangdong Province)
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tumor tissue specimens reveal distinct morphological features of HCC, such as abnormal cell proliferation, altered cellular architecture, and the presence of cancer nests or trabeculae. Pathologists examine these features to confirm the diagnosis, assess the tumor grade and stage, and identify any surrounding normal or precancerous liver tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC group: No previous treatments were performed before MRI examination of patients.
- Non-HCC group: No previous treatments were performed before MRI examination of patients.

SUMMARY:
Abbreviated MRI (AMRI) could improve the diagnostic performance of hepatocellular carcinoma (HCC), but it lacks analysis in different subgroups and effective validation. The investigators aimed to compare and validate the diagnostic performance of different AMRI protocols in diagnosing early-stage HCC.

DETAILED DESCRIPTION:
This retrospective study enrolled untreated patients at risk for developing HCC who underwent gadoxetic acid-enhanced MRI from three independent cohorts from January 2020 to December 2022. Three AMRI protocols were extracted from the complete liver MRI protocol, including non-contrast (NC-AMRI), hepatobiliary phase (HBP-AMRI); and dynamic contrast-enhanced (DCE-AMRI). Two readers at each cohort independently interpreted each AMRI based on ancillary and main features from the Liver Imaging Reporting and Data System (LI-RADS) version 2018. For DCE-AMRI, two established algorithms were employed: modified LI-RADS (DCE-AMRIm) and LI-RADS v2018 (DCE-AMRIv2018). Non-HCCs were ascertained based on histologic and clinical follow-up data, while early-stage HCCs were confirmed post-operatively. Patient-level performance metrics were compared using bootstrap resampling and generalized estimating equations.

ELIGIBILITY:
Inclusion Criteria:

* no previous history of HCC treatment
* no history of any other underlying malignancy besides HCC.

Exclusion Criteria:

* For HCC group: (a) without preoperative MRI within 3 months; (b) without postoperative pathological confirmation; (c) liver cirrhosis without histopathologic proof or radiologic evidence; (d) the size of HCC smaller than 1cm; (e) outside of Milan Criteria; and (f) suboptimal imaging quality.
* For non-HCC group: 1) lost follow-up, 2) insufficient follow-up period, or 3) suboptimal imaging quality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive participants at risk for developing HCC (ie, liver cirrhosis of any etiologies or chronic hepatitis virus infections) who underwent gadoxetic acid-enhanced MRI between January 2020 and December 2022 and are eligible for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 938 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with HCC | immediately after the surgery

SECONDARY OUTCOMES:
Number of patients with non-HCC | immediately after pathology from postoperative or biopsy samples, or clinical diagnosis after at least 1 year without imaging indications of liver malignancy.

CONTACTS AND LOCATIONS:
Locations (1):
- China, Guangdong, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
All data generated for this study are from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Qin Y, Zhang J, Xu D, Zhou X, Ling Z, Li L, Zhao Q, Dong Z, Wang J, Cai HS, Li H, Zhang LG, Feng ST. Diagnosis of Hepatocellular Carcinoma Using Gadoxetic Acid-Enhanced MRI Based on LI-RADS Version 2018 and LI-RADS Modifications. Liver Int. 2025 Nov;45(11):e70366. doi: 10.1111/liv.70366. PMID 41042775